CLINICAL TRIAL: NCT03217292
Title: Evaluation of the Effect of Serratus Anterior Plane Block for Pain Treatment After Video-Assisted Thoracoscopic Surgery
Brief Title: Serratus Anterior Plane Block for Pain Treatment After Video-Assisted Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-KAEK-25 2016/13-06
Record Dates: First submitted 2017-07-02; First posted 2017-07-14 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Nerve Block
MeSH Terms: interventions — Analgesia, Patient-Controlled; Passive Cutaneous Anaphylaxis; Tramadol

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, single-blind
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): IV patient-controlled analgesia (PCA) tramadol+Serratus Anterior Plane Block(SAPB) Tramadol infusion (PCA): 400 mg tramadol, IV 4 mg/mL tramadol solution into 100 mL normal saline; PCA settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
  20 mL of bupivacaine at a concentration of 0.25% to between serratus anterior and intercostal muscle using the in-line technique for SAPB.
  Interventions: Procedure: Serratus Anterior Plane Block; Drug: IV patient-controlled analgesia (PCA) tramadol
- Group T (Active Comparator): IV patient-controlled analgesia (PCA) tramadol Tramadol infusion (PCA): 400 mg tramadol, IV 4 mg/mL tramadol solution into 100 mL normal saline; PCA settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
  Interventions: Drug: IV patient-controlled analgesia (PCA) tramadol

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block
  Arms: Group S
Drug: IV patient-controlled analgesia (PCA) tramadol

SUMMARY:
Analgesia following video-assisted thoracoscopic surgery (VATS) is important for the prevention of postoperative pulmonary complications.Various regional methods of anesthesia are currently being used to achieve this goal. The aim of the study was to assess the effectiveness of SAPB on postoperative VATS analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were in the American Society of Anesthesiologists (ASA) I-III class and underwent video-assisted thoracoscopic surgery (VATS).

Exclusion Criteria:

* Previous history of opioid use preoperatively,
* Allergy to local anesthetics,
* The presence of any systemic infection,
* Uncontrolled arterial hypertension,
* Uncontrolled diabetes mellitus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Postoperative 24 hours
  Visual Analogue Scale was used for pain

SECONDARY OUTCOMES:
tramadol consumption | Postoperative 24 hour
  tramadol consumption
Ramsay sedation scale (RSS) | 24 hours
  Ramsay sedation scale (RSS)

OTHER OUTCOMES:
side effect profile | 24 hours
  side effect profile
additional analgesic use | 24 hours
  additional analgesic use

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Metin Ökmen, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital